CLINICAL TRIAL: NCT04517123
Title: Prone Position and Respiratory Outcomes in Non-Intubated COVID-19 PatiEnts The "PRONE" Study
Acronym: PRONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Duke University (Other); University of North Carolina (Other); University of Miami (Other); University of Pittsburgh (Other); Smith & Nephew, Inc. (Industry); Nox Medical Iceland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00249663
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Pneumonia, Viral
Keywords: covid19; pneumonia; prone positioning; COVID
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Pneumonia | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Usual Care (No Intervention): Usual Care
- Intervention - Prone Positioning (Experimental): Prone Positioning
  Interventions: Other: Prone Positioning

INTERVENTIONS:
Other: Prone Positioning — Prone Positioning
  Arms: Intervention - Prone Positioning

SUMMARY:
The overall objective of this study is to determine whether a positional maneuver (e.g., prone positioning) decreases the need for escalation of respiratory-related care in patients with coronavirus (COVID-19) pneumonia.

DETAILED DESCRIPTION:
As the initial outbreak of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the disease it causes, coronavirus disease 2019 (COVID-19) has spread beyond Wuhan, China it has become a pandemic affecting over 178 countries. Of patients admitted to the ICU, upwards of 85% developed the acute respiratory distress syndrome (ARDS) and most if not all required mechanical ventilation. The beneficial effects of prone positioning for ARDS have been well described. Coupling the reported benefits of prone positioning in COVID-19 associated ARDS patients with the known beneficial effects of early prone-positioning in the treatment of ARDS, it is not surprising that many hospital systems are advocating prone positioning for treatment of ARDS in patients with COVID-19. However, as the pandemic continues to progress in the United States and the number of new cases grows as new clusters emerge, the possibility of 'rationing' ventilators becomes more real. Therefore, therapies that prevent the need for mechanical ventilation are desperately needed. Given the distinct benefit that patients with COVID-19 have with prone positioning, the overarching hypothesis of this trial is that patients with high risk for respiratory failure may also benefit from prone positioning.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* COVID-19 positive by nasopharyngeal swab or serostatus
* Use of supplemental oxygen OR respiratory rate ≥ 20

Exclusion Criteria:

* BMI ≥ 45 kg/m2
* Pregnancy
* Chest tube placement
* Hemodynamic instability with mean arterial pressure < 60 mmHg
* Thoracic or abdominal wounds
* Chest wall deformities
* Vertebral column deformities that would preclude prone positioning
* Facial trauma or surgery in the last 30 days
* Established diagnosis of interstitial lung disease
* Prior single or double lung transplant
* Surgery for spine, femur, or pelvis in the last 3 months
* Thoracic or cardiac surgery in the last 30 days
* Pacemaker placement last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of an escalation in respiratory related care (yes vs no) | During hospitalization, up to 30 days
  Participants will be assessed for the occurrence of an escalation in respiratory related care (Yes or No). Escalation in respiratory related care is clinically defined as any of the following:
  1. intubation
  2. any increase in flow of supplemental oxygen
  3. transition to high flow nasal cannula
  4. increase in fraction of inspired oxygen
  5. transfer from a lower to a higher level acuity of care (e.g. medical floor to intermediate care unit (IMC) or intensive care unit (ICU); IMC to ICU).

SECONDARY OUTCOMES:
Oxygen Saturation | Over a consecutive 24-hour period after randomization
  Oxygen Saturation measured in percent oxygen over a 24-hour period.
Respiratory Effort as assessed by Respiratory Rate | Over a consecutive 24-hour period after randomization
  Respiratory effort will be assessed using the respiratory rate (in breaths per minute) over a 24-hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Punjabi, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Univeristy, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No